CLINICAL TRIAL: NCT00488410
Title: Evaluation of the Forecasts Parameters of Real Time Three-dimensional Doppler Echocardiography in Selecting Patients With Chronic Heart Failure for Cardiac Resynchronisation Therapy
Brief Title: SYNCHRO. Evaluation of the Forecasts Parameters of Real Time-three-dimensional Doppler Echocardiography in Selecting Patients With Chronic Heart Failure for Cardiac Resynchronisation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: CHU Clermont-Ferrand, Cardiac surgery center
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: CHU63-0016
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Heart Failure
Keywords: Chronic heart failure; real time three-dimensional echocardiography; cardiac resynchronization therapy; ventricular asynchrony; systolic dysynchrony index
MeSH Terms: interventions — Echocardiography, Doppler

INTERVENTIONS:
Device: Doppler echocardiography

SUMMARY:
Patients showing a normal value of SDI (< or + 8%) will randomly be assigned to CRT in "ON" or "OFF"mode at one month after implantation. In any case of emergency, an automated rescue mode is included in the device for the patients in "OFF" mode.

DETAILED DESCRIPTION:
Patients with a pathological SDI (> 8%) will as usually be treated by CRT and will serve as control group. The study duration for each patient included in the trial is 6 months. Patients showing a decreased NYHA score by at least one class and an absence of major cardiovascular event during the period will be considered as "good responders". The otherswill be considered as "no responders".

Based on this composite clinical score, the percentage of good responders in each group at 6 months is the primary endpoint of the study.

Main secondary endpoints :

* Evaluation of the left ventricular function
* Exercice capacity
* Serious adverse events'frequency
* Quality of life (SF36)
* Diagnostic and prognostic value of the "Brain Natriuretic Peptide"(NT pro BNP)evolution.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Age>18 years
* Patients in functional class NYHA III or IV
* Patient with ejection fraction <or=150msec or with QRS between 120 and 149 msec but with echocardiographic evidences for cardiac dyssynchrony, such as those retained in the CARE-HF trial, e.g.two from the three following criterions :-Aortic pre-ejection delay>140msec
* Interventricular mechanical delay >40msec
* Delayed activation of the left ventricular postero-lateral wall
* Patient under optimal treatment for chronic heart failure for at least one month before inclusion
* Written informed consentement

Exclusion Criteria:

* Patient with atrial fibrillation
* Absence of echogenicity
* Patient with an indication for pacemaker implantation
* Patient suffering from arterial pressure disorders, with systolic pressure greater than 170 or lower than 80 mmHg
* Major cardiovascular event within 6 weeks before inclusion
* Patient in the exclusion period of any other clinical trial
* Patient without social insurance policy
* Drug or alcohol addiction
* Any psychological disorder
* Pregnant women
* Patient with a transplanted organ
* HIV positive serology at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-11; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Three parallel arms, randomized, controlled, single blinded, monocentre, clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Citron, Pr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France